CLINICAL TRIAL: NCT06271902
Title: Effects of the Singapore Youth Shoulder Overuse Injury Prevention Program (YoSO-IPP) Among Youth Volleyball Athletes in Singapore: a Randomized Controlled Trial
Brief Title: Effects of the Singapore Youth Shoulder Overuse Injury Prevention Program Among Youth Volleyball Athletes in Singapore
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, swarup mukherjee, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2023-531
Record Dates: First submitted 2024-02-02; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Sport Injury

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with an intervention group and a control group to evaluate the effects of the YoSO-IPP. The intervention group will perform the exercises and attend the online educational workshop. The control group will only perform lower body stretching exercises which is considered as a sham program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will be instructed to perform YoSO-IPP at a recommended frequency of two times per week for 12 weeks and attend an online 45-minute educational workshop in Week 1
  Interventions: Other: Singapore Youth Shoulder Overuse Injury Prevention Program
- Control group (Active Comparator): Participants will be instructed to perform the lower body stretching program at a recommended frequency of two times per week.
  Interventions: Other: Lower body stretching program

INTERVENTIONS:
Other: Singapore Youth Shoulder Overuse Injury Prevention Program — A 10-minute, 4-exercises program that targets shoulder eccentric external rotation strength, shoulder internal rotation range of morion, and thoracic rotation range of motion. The topic for the 45-minute educational workshop will be on overuse injuries among youth athletes.
  Arms: Intervention group
Other: Lower body stretching program — A 10-minute, 5-stretches sham exercise program that does not target the upper extremity and are only held for 10 seconds.
  Arms: Control group

SUMMARY:
The Singapore Youth Shoulder Overuse Injury Prevention Program (YoSO-IPP) includes an exercise segment and an education segment. This study will (1) assess the effects of the exercise segment, and (2) assess the effects of the education segment among youth volleyball athletes using a randomized controlled trial over 12 weeks. Performance outcome measures of shoulder eccentric external rotation strength, shoulder internal rotation range of motion, and thoracic rotation range of motion will be used to assess the effects of the exercise segment. Knowledge scores via an online questionnaire will be used to assess the effects of the education segment.

Hypothesis: The YoSO-IPP will have an effect on shoulder eccentric external rotation strength, shoulder internal rotation range of motion, and thoracic rotation range of motion and on knowledge scores.

DETAILED DESCRIPTION:
A randomized controlled trial study design will be utilized to assess the effects of YoSO-IPP over 12 weeks. A within-team randomization will be conducted. This is to ensure a good balance between the intervention and control groups as different teams have different training regimes, training frequencies and training intensities.

Participants in the intervention group will be required to perform the exercise segment of YoSO-IPP for 12 weeks, at a recommended frequency of two times per week - (a) cross-body stretch, (b) eccentric external rotation shoulder strength exercise, (c) trunk rotation, and (d) modified cat-cow thoracic mobility exercise.

Participants in the control group will be required to perform lower body stretches for 12 weeks, at a recommended frequency of two times per week - (a) double leg calf stretch, (b) quadriceps stretch, (c) hip flexor stretch, (d) seated single leg hamstring stretch, and (e) seated single gluteal stretch. This stretching program is considered a sham program in this study as it does not target the upper extremity and the stretches are only held for 10 seconds.

Participants in both groups will each receive an instruction booklet for their respective program. Respective instructional videos will also be distributed. For the following 12 weeks, participants are to perform the exercises at a recommended frequency of two times per week. They will also be required to report the number of times they performed their respective programs that week via an online questionnaire weekly.

Participants who are randomized into the intervention group will attend an online 45-minute educational workshop in Week 1. This is the education segment of YoSO-IPP. Participants who are randomized into the control group will not attend the online 45-minute educational workshop.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years old youth athlete; in the sport of volleyball; trains with an aim to compete; currently NOT undergoing any shoulder or elbow overuse injury prevention program

Exclusion Criteria:

* Below 12 and above 18 years old; not in the sport of volleyball; trains without an aim to compete; currently undergoing a shoulder or elbow overuse injury prevention program

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Shoulder external rotation strength | Baseline (Week 0), Week 6, Week 12
  Shoulder external rotation strength is a performance outcome measure of interest. It will be measured using a handheld electronic dynamometer. It will be presented in Newtons (N).
Internal rotation range of motion | Baseline (Week 0), Week 6, Week 12
  Shoulder internal rotation range of motion is a performance outcome measure of interest. It will be measured using 'Clinometer', a validated phone application for range of motion measurement. It will be presented in degrees (°).
Thoracic rotation range of motion | Baseline (Week 0), Week 6, Week 12
  Thoracic rotation range of motion is a performance outcome measure of interest. It will be measured using 'Clinometer', a validated phone application for range of motion measurement. It will be presented in degrees (°).
Knowledge of overuse injuries | Baseline (Week 0), Week 12
  Knowledge scores will be calculated based on a novel questionnaire concerning youth athletes and overuse injuries. The scores will range from 0 to 20, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Shoulder overuse injury prevalence | Baseline (Week 0), Week 12
  Injury prevalence will be determined based on the Youth Overuse Injury Questionnaire (YOvIQ).
Elbow overuse injury prevalence | Baseline (Week 0), Week 12
  Injury prevalence will be determined based on the Youth Overuse Injury Questionnaire (YOvIQ).
Shoulder overuse injury severity | Baseline (Week 0), Week 12
  Injury severity will be determined based on the Youth Overuse Injury Questionnaire (YOvIQ). Severity score will range from 0 to 100, with higher scores indicating a more severe injury.
Elbow overuse injury severity | Baseline (Week 0), Week 12
  Injury severity will be determined based on the Youth Overuse Injury Questionnaire (YOvIQ). Severity score will range from 0 to 100, with higher scores indicating a more severe injury.

CONTACTS AND LOCATIONS:
Overall Officials: Mukherjee, Principal Investigator — Nanyang Technological University, National Institute of Education
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be available upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. End 5 years.
Access Criteria: Access subject to approval by Principal Investigator.

REFERENCES:
- [Background] Lau R, Mukherjee S. Prevalence of Shoulder and Elbow Overuse Injuries Among Competitive Overhead Youth Athletes in Singapore. Orthop J Sports Med. 2023 Mar 21;11(3):23259671231156199. doi: 10.1177/23259671231156199. eCollection 2023 Mar. PMID 36970317
- [Background] Lau R, Mukherjee S. Developing the Singapore youth shoulder overuse injury prevention program. Phys Ther Sport. 2024 Jan;65:30-37. doi: 10.1016/j.ptsp.2023.11.001. Epub 2023 Nov 16. PMID 38006797